CLINICAL TRIAL: NCT01182636
Title: A Randomized, Double-Blind, Multiple-Site, Placebo Controlled, Parallel Design, Clinical Study to Evaluate the Bioequivalence of Adapalene Gel 0.1% (PLIVA Research & Development Ltd.) Compared to Differin® (Adapalene 0.1%) Topical Gel (Galderma Laboratories) in Patients With Acne Vulgaris
Brief Title: Bioequivalence of Adapalene Topical Gel in Patients With Acne Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 70716202
Record Dates: First submitted 2010-08-13; First posted 2010-08-17 (Estimated); Last update posted 2010-11-24 (Estimated); Status verified 2010-11

CONDITIONS: Acne Vulgaris
Keywords: Bioequivalence; Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Investigational Test Product (Experimental): Adapalene Topical Gel, 0.1%
  Interventions: Drug: Adapalene
- Reference Listed Drug (Active Comparator): Differin® (adapalene 0.1%) Topical Gel
  Interventions: Drug: Differin®
- Placebo (Placebo Comparator): Gel base only
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Adapalene — 0.1% Topical Gel
  Arms: Investigational Test Product
Drug: Differin® — 0.1% Topical Gel
  Other Names: Adapalene
  Arms: Reference Listed Drug
Drug: Placebo — Gel Base
  Arms: Placebo

SUMMARY:
The objective of this study was to evaluate the efficacy and safety of the test formulation of adapalene gel 0.1% (PLIVA Research & Development Ltd.) as compared to the already marketed formulation, Differin® (adapalene 0.1%) topical gel (Galderma Laboratories) in patients with acne vulgaris.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria for Comparative Clinical Endpoint Studies.

Statistical Methods: FDA Bioequivalence Statistical Methods for Comparative Clinical Endpoint Studies.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating female, 12-40 years of age inclusive.
* Signed informed consent form, which meets all the criteria of the current FDA regulations. For patients under the age of majority in the state they are enrolled, the patient's parent or legal guardian will be required to sign the consent form and the patient will sign an IRB approved "assent to participate" form.
* If female and of child bearing potential, prepare to abstain from sexual intercourse or use reliable method of contraception during the study (i.e. condom, Intrauterine device, hormonal contraceptives). Patients on hormonal contraceptives must have been on the same hormonal contraceptive for 3 months prior to the baseline visit and continue throughout the duration of the study.
* Have moderate to severe facial acne as defines as: at least 20 but no more that 60 facial inflammatory lesions (papules and pustules) and at least 25 but no more than 100 non-inflamed lesions (open and closed comedones) and have a Physician's Global Assessment score of 3, 4, or 5.

Exclusion Criteria:

* Patient has more than 2 facial nodular lesions, any nodules present will be documented but will not be included in the inflammatory lesion count.
* Patient has active cystic acne.
* Patient has acne conglobate.
* Patient with significant facial hair such as beards or tattoos or excessive facial scarring that, in the Investigator's opinion, may interfere with the evaluation of the patient's acne.
* Patients with facial sunburn.
* Any dermatological condition other than acne vulgaris that, in the Investigator's opinion, may interfere with the evaluation of the patient's acne (e.g. rosacea, psoriasis, dermatitis).
* Females who are pregnant, lactating, or likely to become pregnant during the study.
* History of allergy or sensitivity to adapalene or other retinoids, or history of any drug hypersensitivity or intolerance which, in the Investigator's opinion, would compromise the safety of the patient or the study.
* Significant history or current evidence of chronic infectious disease, system disorder, organ disorder, or other medical condition that, in the Investigator's opinion, would place the study participant at undue risk by participation.
* Use of any topical antibiotics, topical steroids, or topical anti-inflammatory products used on the face, any oral antibiotics known to treat acne, any systemic steroids, or any systemic anti-inflammatory agents (other than the use of non-steroidal anti-inflammatory agents) within 28 days of the first dosing day.
* Use of oral isotretinoin (Accutane®) within 6 months. Use of topical tretinoin (Retin-A®), adapalene (Differin®), tazarotene (Tazorac®), or azelaic acid (Azelex®) within 28 days of the first dosing day.
* Receipt of any drug as part of a research study within 30 days prior to dosing.
* Female patients who are using hormonal contraceptives must have been on the same type and strength of hormonal contraceptive for at least 3 months prior to enrollment in the study and throughout the duration of the study.
* Patients should not use any medicated facial products (soaps, lotions, moisturizers, etc.) or other medicated facial cleansing agents for 14 days prior to study enrollment.
* Previous participation in this study.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 601 (Actual)
Dates: Start 2007-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Mean Percent Reduction from Baseline in Non-Nodular Inflamed Lesion Count | 84 days
  Per Protocol Population (PPP) was assessed for the mean percent reduction compared to baseline in non-nodular lesion count (papules and pustules) at Day 84. If a patient was withdrawn from the study prior to Day 84 for lack of efficacy, then their data was carried forward for this analysis.
Mean Percent Reduction from Baseline in Non-Inflamed Lesion Count | 84 days
  Per Protocol Population (PPP) was assessed for the mean percent reduction in non-inflamed lesion count (open and closed comedones) compared with baseline at Day 84. If a patient was withdrawn from the study prior to Day 84 for lack of efficacy, then their data was carried forward for this analysis.
Safety Analysis | 84 Days
  All 601 patients randomized and dispensed study drug were included in the safety analysis. The frequency, severity, and relationship to the study drug for adverse events in each treatment group were used to compare the safety of the study medications.

SECONDARY OUTCOMES:
Mean Numerical Reduction in Inflamed Lesion Counts | 84 Days
  Secondary measure of bioequivalence using the Intent-to-Treat (ITT) population.
Mean Numerical Reduction in Non-Inflamed Lesion Counts | 84 Days
  Secondary measure of bioequivalence using the Intent-to-Treat (ITT) population.
Proportion of Patients Considered a "Clinical Success" or "Clinical Failure" | 84 Days
  Secondary measure of bioequivalence using the Intent-to-Treat (ITT) population. "Clinial Success" or "Clinical Failure" is defined by the Physician's Global Assessment.

CONTACTS AND LOCATIONS:
Locations (21):
- United States (19):
  - Dermatology Research of Arkansas, Little Rock, Arkansas
  - Dermatology Research Associates, Los Angeles, California
  - Cherry Creek Research, Inc., Denver, Colorado
  - University Clinical Research, Inc., Pembroke Pines, Florida
  - MedaPhase, Inc., Newnan, Georgia
  - SNBL Clinical Pharmacology Center, Inc., Baltimore, Maryland
  - Michigan Center for Research Corportation, Clinton Township, Michigan
  - Office of Atoya Breona Adams, MD, Las Vegas, Nevada
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Helendale Dermatology & Medical Spa, LLC, Rochester, New York
  - Dermatology Associates of Rochester, PC, Rochester, New York
  - Office of Zoe Diana Draelos, MD, High Point, North Carolina
  - University Dermatology Consultants, Inc., Cincinnati, Ohio
  - Novum Pharmaceutical Research Services, Pittsburgh, Pennsylvania
  - Knoxville Dermatology, PC, Knoxville, Tennessee
  - Arlington Center for Dermatology, Arlington, Texas
  - Center for Clinical Studies, Houston, Texas
  - Dermatology Associates of Tyler, Tyler, Texas
  - Aurora Advanced Healthcare, Inc., Milwaukee, Wisconsin
- Belize (2):
  - Dermatology and Skin Surgery Centre, Belize City
  - FXM Research International, Belize City